CLINICAL TRIAL: NCT03854565
Title: Predictive Value of Glycocalyx Biomarkers in Mechanical Ventilation of Patients With ARDS for Clinical Prognosis and Long-term Pulmonary Fibrosis
Brief Title: Glycocalyx Biomarkers in ARDS for Clinical Prognosis and Pulmonary Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Chun Pan, Principal Investigator, Southeast University, China
Other Study IDs: Decorin-ARDS fibrosis study
Record Dates: First submitted 2019-02-17; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: ARDS, Human; Endothelial Dysfunction; Mechanical Ventilation Pressure High
Keywords: ARDS; Endothelial Dysfunction; mechanical ventilation; Glycocalyx; pulmonary fibrosis; mortality
MeSH Terms: conditions — Respiratory Distress Syndrome; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — blood and urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild ARDS: patients have mild ARDS according to Berlin definition
  Interventions: Diagnostic Test: Glycocalyx measurement，respiratory mechanics measurement
- Moderate ARDS: patients have moderate ARDS according to Berlin definition
  Interventions: Diagnostic Test: Glycocalyx measurement，respiratory mechanics measurement
- Severe ARDS: patients have severe ARDS according to Berlin definition
  Interventions: Diagnostic Test: Glycocalyx measurement，respiratory mechanics measurement

INTERVENTIONS:
Diagnostic Test: Glycocalyx measurement，respiratory mechanics measurement — ELASA measure glycocalyx, measure plateau pressure, driving pressure

SUMMARY:
ARDS is a severe disease in ICU, and could induce high mortality. Glycocalyx is an important matrix construction which covers endothelial cells, it could protect endothelial cells injury and the glycocalyx biomarkers could predict pulmonary injury.

Decorin is a member of the small leucine-rich proteoglycan (SLRP) family, contains a single glycosaminoglycan (GAG) chain and a core protein with 12 leucine-rich repeats. In the previous study, decorin is associated with cardiac and liver fibrosis, however, the effects of decorin on ARDS pulmonary fibrosis have not been clarified.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18yrs and <80yrs
2. Meet ARDS Berlin definition
3. With mechanical ventilation

Exclusion Criteria:

1. have chronic pulmonary disease
2. have use heparin or low molecular heparin or chondroitin sulfuric acid

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients have been diagnosed ARDS with mechanical ventilation, and do not been used heparin, molecular heparin, chondroitin sulfuric acid.
Sampling Method: Probability Sample
Enrollment: 336 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
28 days mortality from patients involved in the study | 28 days
  28 days mortality from patients involved in the study

SECONDARY OUTCOMES:
CT and syndecan-1 to evaluate pulmonary fibrosis | 1mon, 3mon and 6 month
  pulmonary fibrosis evaluated by biomarker and CT
pulmonary function test to evaluate pulmonary function | 1mon, 3mon and 6 month
  pulmonary function evaluated by pulmonary function test

CONTACTS AND LOCATIONS:
Overall Officials: Chun C Pan, Dr, Principal Investigator — Zhongda hospital, Southeast University, Jiangsu, China
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided